CLINICAL TRIAL: NCT06612528
Title: Effect of Transcranial Direct Current Stimulation on Singers' Voice
Brief Title: Transcranial Direct Current Stimulation on Singer's Voice
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Phd, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5.758.856
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Voice; Voice Range Profile; Voice Quality
Keywords: transcranial direct current stimulation; tDCS; Flexible tube; voice; singers
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Hydrotherapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three groups (M1, Cerebellum, or sham) using a computer-generated randomization list. All participants will receive 10 consecutive sessions of anodal tDCS combined with vocal exercises, except on weekends. Stimulation parameters and electrode placement varied by group: M1 - C5 (anode) and contralateral supraorbital (cathode); Cerebellum - cerebellar cortex (anode) and right deltoid (cathode); sham - identical electrode placement to the Cerebellum group, but with stimulation ceasing 30 seconds after onset. Vocal exercises consisted of four 3-minute bouts with a 2-minute rest between bouts. To maintain blinding, a towel was placed over the participant&amp;#39;s head during the procedure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- M1 and vocal exercise (Experimental): anodal tDCS over primary motor cortex associated with the vocal exercise using the flexible tube in water.
  Interventions: Device: tDCS; Device: Flexible tube in water
- Cerebellum and vocal exercise (Active Comparator): anodal tDCS over cerebellum associated with the vocal exercise using the flexible tube in water.
  Interventions: Device: tDCS; Device: Flexible tube in water
- Sham and vocal exercise (Placebo Comparator): tDCS sham associated with the vocal exercise using the flexible tube in water.
  Interventions: Device: tDCS; Device: Flexible tube in water

INTERVENTIONS:
Device: tDCS — The tDCS is a non-invasive brain stimulation technique. In this study, we used an intensity of 2mA for 20 minutes in two different areas.
  M1 group: the anode was over C5 (10-10 EEG system) and the cathode was placed over Fp2. For the Cerebellum group stimulation, the targeted anode area was 2 cm below the inion and the cathode over the deltoid muscle.
  Other Names: transcranial direct current stimulation
Device: Flexible tube in water — The exercise involved producing sustained /u/ vowels in ascending and descending scales, tailored to each participants vocal range.
  The flexible tube was 35 cm long, 1 cm in diameter, and 2 mm thick. One end of the tube was submerged 3 cm into a 500 ml bottle filled with water. Participants produced four sets of vocal exercises, each lasting 3 minutes, with 2-minute rests between sets, totaling 20 minutes of vocal therapy.
  Other Names: Lax vox; Flexible tube

SUMMARY:
Transcranial direct current stimulation (tDCS) can be used to temporarily and reversibly modulate brain functions and is an increasingly utilized tool to investigate the relationships between brain and behavior. This study aimed to identify the effects of tDCS on vocal quality, vocal range, neuromotor functioning of the larynx and self-reported vocal effort in vocally healthy singers. This is a triple-blinded, sham-controlled, randomized clinical trial. The participants will be randomized to one of the three tDCS groups (primary motor cortex, cerebellum or sham). In each group a voice training will be applied at the same tDCS time. The three groups are: (i) cerebellum; (ii) primary motor cortex (M1); (iii) sham. The tDCS parameters in the active groups are anodal - 2mA for 20 minutes, at the sham group the stimuli are finished 30 secondes before starting. Volunteers will pass for 10 intervention days and they will be evaluated for vocal performance before the sessions, in the day 5 of intervention, the last day of intervention (day 10) and 1 month later for follow up evaluation. Voice recordings will be take to assess the following vocal parameters: vocal range profile (VRP) at weak and strong intensities; vocal quality (jitter, shimmer, irregularity, glottal-to-noise excitation ratio, and dysphonia acoustic index) at weak, habitual, and strong intensities; laryngeal diadochokinesis, and self-reported vocal effort using the adapted Borg CR10 scale.

DETAILED DESCRIPTION:
Data collection is being conducted at the Applied Neuroscience Laboratory (LANA) of the Federal University of Pernambuco (UFPE). Videolaryngoscopy is performed at the UFPE Hospital, in the laryngology outpatient clinic.

This phase of the study includes vocally healthy individuals who are singers without formal music or singing training. Residents of the city of Recife and the Metropolitan Region, aged 18 to 45 years. The age range was chosen considering the period of maximum vocal efficiency To determine the sample size, in phase 2, a pilot study was conducted with 15 participants that will serve as a parameter for sample size calculation. This will be done using the G*Power 3.1 program, considering a statistical power (β) of 80% and a significance level (α) of 5%. For this analysis, the primary vocal outcome variables (vocal range profile) will be considered, and the sample size will be considered the largest value among the selected outcomes.

Singers without formal music training and without vocal complaints are included. In order to assess vocal health, all singers underwent videolaryngoscopy, performed by an otolaryngologist. After the exam, subjects are selected who, according to the otolaryngologist's report, presented functional anatomical and physiological conditions. Individuals with minimal structural alterations (MSA) will not be excluded, as long as the glottal closure is complete and with regular glottal vibration on stroboscopy.

Individuals who are smokers or who present signs and symptoms of laryngeal, pharyngeal or respiratory diseases at the time of data collection are excluded from the sample. Volunteers who use neuroactive medications regularly, have metal implants in the cervical region or above, and have any history of seizures or epilepsy will also be excluded.

The sample of singers is being constituted by convenience through individuals who are singers without vocal complaints of both sexes, recruited through advertisements in electronic media. The first contact with the volunteers is through a screening to verify the eligibility criteria.

The same data collection instruments from phase 1 are used in phase 2 of this study. Added to this is the vocal exercise, performed with the aid of a silicone tube with the following dimensions: 35cm in length, 1cm in diameter and 2mm in thickness, and with the distal end immersed at a distance of 3cm from the bottom of a 500ml plastic bottle containing 2/3 of water and with the spaces delimited. This study seeks to investigate the combined effects of tDCS and vocal exercises on singers' voices. We will conduct a clinical trial to examine the impact of concurrent neuromodulation and vocal training. Anodal tDCS will be applied at 2mA for 20 minutes to three groups: (i) M1; (ii) Cerebellum; and (iii) sham. All groups will also perform vocal exercises using a flexible tube (FT) for a total of 12 minutes. Participants will complete an adverse effects questionnaire after each session to report any discomfort. Vocal assessment is performed before the intervention to obtain results on vocal parameters, vocal range profile, and vocal effort, as well as on the 5th day after the start of the intervention, on the 10th day, and 1 month after the end of the activities. The entire assessment procedure is being performed as described in phase 1 of this study, only the request for the vocal task to assess perceived effort is different in the phase 2 singers. In this case, the participants answered the same Borg CR 10-BR scale questionnaire - adapted for vocal effort to assess the singers' self-perception of the proposed tasks, however, the singers are instructed to report the intensity of the effort produced during the singing task of a song of their choice, according to their self-perceived difficulty.

In order to determine the volunteers who would be in each group, and for subsequent sample size calculation, a randomization was performed for 15 volunteers, by an external researcher, using a random table and adjusted to allow for counterbalancing Codes were assigned to the groups, which were kept in opaque and numbered envelopes, available only to the person responsible for applying the tDCS. In this way, the evaluator, the therapist responsible for the vocal technique with a flexible tube immersed in water, and the singer remain "blind" to the type of stimulation to which the participants are subjected. After performing the sample size calculation, a new randomization will be performed to allocate the participants who will continue in the data collection to complete the number of necessary volunteers.

The participants are allocated into three groups, namely: (i) M1; (ii) Cerebellum; (ii) sham. In all groups, 10 consecutive sessions of anodal tDCS associated with vocal exercise are performed, these only do not occur on weekends. For the application of tDCS in the groups: (i) M1, the stimulation electrode (anode) is positioned over C5 (international 10-20 EEG system) with the cathode (negative pole) positioned over the contralateral supraorbital region; (ii) Cerebellum, the stimulation electrode over the cerebellar cortex (inion, slightly to the right) and the reference electrode (cathode) is positioned over the right deltoid muscle; (ii) sham, the montage equivalent to cerebellar stimulation is performed, however in the sham stimulation there is an interruption of the stimulation 30 seconds after the start, thus the current intensity drops to zero mA, but the electrodes remained on the scalp of the volunteers until the end of the vocal exercise. The exercise with FT is performed for a total of 20 minutes (3 minutes of FT, four sequences, followed by 2 minutes of interval) in all groups. In the sham group, the electrodes are only removed after the end of the vocal exercises, so that the patient is unaware of the type of stimulation (real or sham) to which they were exposed. To blind the evaluator and therapist, a towel is placed over the volunteer's head every day. Participants were instructed to sit comfortably while electrodes were placed on their scalp and tDCS stimulation was initiated. Following stimulation, participants performed vocal exercises using a flexible tube. The exercise involved producing sustained /u/ vowels in ascending and descending scales, tailored to each participant's vocal range (soprano, mezzo-soprano, contralto, tenor, baritone, or bass). These scales were based on pre-recorded piano accompaniments.

The flexible tube was 35 cm long, 1 cm in diameter, and 2 mm thick. One end of the tube was submerged 3 cm into a 500 ml bottle filled with water. Participants produced four sets of vocal exercises, each lasting 3 minutes, with 2-minute rests between sets, totaling 20 minutes of vocal therapy. This ensured that the vocal exercises concluded simultaneously with the tDCS session. Voice recordings will be take to assess the following vocal parameters: vocal range profile (VRP) at weak and strong intensities; vocal quality (jitter, shimmer, irregularity, glottal-to-noise excitation ratio, and dysphonia acoustic index) at weak, habitual, and strong intensities; laryngeal diadochokinesis, and self-reported vocal effort using the adapted Borg CR10 scale. This research was conducted in accordance with the ethical guidelines established by Brazil's National Health Council (Resolution 466/12). The study was approved by the Human Research Ethics Committee of UFPE's Health Sciences Center (number 5.758.856). Participants provided written informed consent after being fully informed about the study's objectives, procedures, potential risks, and benefits.

While the study posed minimal risks, participants might experience mild side effects from tDCS, such as tingling, itching, or burning sensations at the electrode sites. These side effects were carefully monitored. Additionally, some participants might experience discomfort during videolaryngoscopy or vocal exercises. However, these issues were addressed promptly.

Participants benefited from receiving guidance on vocal health and a personalized flexible tube. Data collected from vocal assessment software will be stored securely for at least 5 years. All data collected using Vocalgrama and VoxMetria software were analyzed using the respective software. In Vocalgrama, the following outcome measures were extracted: minimum and maximum fundamental frequency (f0), f0 range, st range, minimum and maximum intensity, and area of the vocal range profile. In VoxMetria, the following measures were extracted: jitter, shimmer, noise-to-harmonic ratio (NHR), and average perturbation quotient (APQ) from a 6-second sustained /ε/ vowel, excluding the first and last seconds. Audio recordings were made at a sampling rate of 44 kHz and 16-bit resolution. VoxMetria was also used to count the number of peaks in diadochokinetic tasks. Perceived effort was assessed using the Borg CR 10-BR scale adapted for vocal effort.

Data normality will be assessed using the Shapiro-Wilk test. The ANOVA repeated mensures will be applied between the times of evaluation. All analyses will be performed using SPSS (version 26.0, SPSS Inc, Chicago, USA) with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Vocally healthy singers without formal singing education

Exclusion Criteria:

* Participants will be excluded from the sample if they were smokers, had abnormalities in previous otorhinolaryngological examination, or exhibited signs and symptoms of laryngeal, pharyngeal, or respiratory diseases at the time of collection. Volunteers who regularly used neuroactive medications, had metallic implants in the cervical region or above, or had any history of seizures or epilepsy will also be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Vocal Range Profile | From enrollment to the end of evaluation at 6 weeks
  Minimum fundamental frequency - f0; Maximum f0; Extension f0; Extension in Semitone; Minimum intensity; Maximum intensity and Area

SECONDARY OUTCOMES:
Vocal quality | From enrollment to the end of evaluation at 6 weeks
  jitter, shimmer, irregularity, Glottal-to-noise-excitation ratio, Dysphonia Acoustic Index

OTHER OUTCOMES:
Larynx neuromuscular control and coordination | From enrollment to the end of evaluation at 6 weeks
  Diadochokinesis of the larynx
Self-reported vocal effort | From enrollment to the end of evaluation at 6 weeks
  Using the Adapted Borg CR10 for Vocal Effort Ratings (BR), maintained a scale from 0 to 10, where 0 means "no vocal effort at all", and 10 "maximum vocal effort"

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil